CLINICAL TRIAL: NCT01317303
Title: Comparison of Measures of Plasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UNSW10106
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Depression; Healthy
Keywords: paired associative stimulation; theta burst stimulation; transcranial magnetic stimulation; neuroplasticity; healthy controls
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PAS25 (Experimental): PAS25 refers to the intervention 'paired-associative stimulation' with peripheral ulnar nerve stimulation followed by TMS to the motor cortex 25 ms after.
  Interventions: Procedure: PAS25
- cTBS-PAS (Experimental): 40 seconds of continuous Theta-burst stimulation, followed by PAS25 which refers to the intervention 'paired-associative stimulation' with peripheral ulnar nerve stimulation followed by TMS to the motor cortex 25 ms after.
  Interventions: Procedure: cTBS-PAS25
- iTBS (Experimental): 190 seconds of intermittent theta-burst stimulation
  Interventions: Procedure: iTBS
- cTBS-iTBS (Experimental): 40 seconds of continuous Theta-burst stimulation, followed by 190 seconds of intermittent Theta-burst stimulation
  Interventions: Procedure: cTBS-iTBS

INTERVENTIONS:
Procedure: cTBS-PAS25 — 40 seconds of continuous Theta-burst stimulation, followed by PAS25 which refers to the intervention 'paired-associative stimulation' with peripheral ulnar nerve stimulation followed by TMS to the motor cortex 25 ms after
  Other Names: Magstim,; Digitimer
  Arms: cTBS-PAS
Procedure: cTBS-iTBS — 40 seconds of continuous Theta-burst stimulation, followed by 190 seconds of intermittent Theta-burst stimulation
  Arms: cTBS-iTBS
Procedure: PAS25 — PAS25 refers to the intervention 'paired-associative stimulation' with peripheral ulnar nerve stimulation followed by TMS to the motor cortex 25 ms after.
  Other Names: Magstim; Digitimer
  Arms: PAS25
Procedure: iTBS — 190 seconds of intermittent theta-burst stimulation
  Other Names: Magstim
  Arms: iTBS

SUMMARY:
Neuroplasticity refers to the ability of the nerve cells to modify their structure or function in response to injury or insult, or other environmental stimuli, with these changes outlasting the period of exposure. Plasticity may be observed as short term or long term changes. In humans, neuroplasticity can be readily assessed in the motor cortex, as excitability changes are demonstrated in the degree to which peripheral muscles are activated, seen through changes in motor-evoked potentials (MEPs). In this study, a number of approaches to assessing neuroplasticity will be evaluated: Paired-associative stimulation (PAS), Theta Burst Stimulation (TBS), which is a form of transcranial magnetic stimulation (TMS) and protocols that combine these two. In addition, participants will complete a computerised 'rotor pursuit task' designed to provide a measure of motor learning.

The investigators aim to find the most efficacious (defined by greatest number of responders and effect size as seen in an increase in MEP amplitude) brain stimulation protocol. The investigators will expose the same participants to four excitatory conditioning stimulation paradigms, with each session separated by at least a week.

Our hypotheses include:

The four conditioning stimulation protocols should increase motor cortical excitability, the investigators therefore expect there to be a significant increase in participant MEPs, with a positive correlation in the increase ofMEP amplitude of the protocols. The investigators do however expect that due to the principles of homeostatic metaplasticity, that the protocols preceded by cTBS will show greater MEP change, due to the lowering of the threshold for LTP plasticity induction. In addition, the investigators expect that an increase in the motor learning manifest by the rotor pursuit task and for there to be a correlation in participants between the increase in MEP amplitude and the improvement in time on target (TOT) shown in the motor learning task (MLT).

ELIGIBILITY:
Inclusion Criteria:

* healthy controls
* those suffering depression
* aged

Exclusion Criteria:

1. Significant Neurological illness, including epilepsy
2. Alcohol use above NHRMC guidelines
3. Illicit drug use
4. Electronic implant; such as cochlear implant or pacemaker
5. Musculoskeletal disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
amplitude of motor evoked potentials | 60 minutes post brain stimulation protocol intervention

SECONDARY OUTCOMES:
motor learning through performance on a 'rotor pursuit task' | time frame relates to 5 blocks of 5 trials for each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute, University of New South Wales, Sydney, New South Wales, Australia

REFERENCES:
- See also: Black Dog Institute website — http://www.blackdoginstitute.org.au